CLINICAL TRIAL: NCT02131870
Title: Study of the Iron Absorption From Capsules Containing Lactobacilli and Iron
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Probi AB (Industry)
Responsible Party: Sponsor
Model: Crossover | Purpose: Basic Science
Other Study IDs: ProIron
Record Dates: First submitted 2014-04-30; First posted 2014-05-06 (Estimated); Last update posted 2014-08-15 (Estimated); Status verified 2014-08

CONDITIONS: Healthy
Keywords: iron absorption; healthy females; child bearing age

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- L plantarum DSM 9843 (Active Comparator)
  Interventions: Dietary Supplement: L plantarum DSM 9843 or placebo
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: L plantarum DSM 9843 or placebo

INTERVENTIONS:
Dietary Supplement: L plantarum DSM 9843 or placebo

SUMMARY:
The purpose of this study is to study the effect of a probiotic product on iron absorption in healthy females of child-bearing age.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Age ≥19 and ≤45 years
* Hb >117g/L

Exclusion Criteria:

* Gastrointestinal diseases
* Metabolic diseases
* Use of other probiotic products during the study and 2 weeks before the study start
* Pregnant or breast-feeding
* A serum ferritin level >60 µg/L
* Medication (oral contraceptives allowed)
* Intake of dietary supplements (incl. iron) during the study and two weeks before the study start
* No blood donation in the last 2 months
* High C-reactive protein levels

Ages: 19 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Dates: Primary Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Iron absorption ratio in blood samples | 14 days
  Iron absorption will be estimated by measuring the isotope ratio (55Fe/59Fe) in blood after addition of iron isotopes in test meals (55Fe in placebo meal, 59Fe in L plantarum DSM 9843 meal).

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Internal Medicin and Clinical Nutrition, the Sahlgrenska Academy, Gothenburg University, Gothenburg, Sweden

REFERENCES:
- [Derived] Hoppe M, Onning G, Hulthen L. Freeze-dried Lactobacillus plantarum 299v increases iron absorption in young females-Double isotope sequential single-blind studies in menstruating women. PLoS One. 2017 Dec 13;12(12):e0189141. doi: 10.1371/journal.pone.0189141. eCollection 2017. PMID 29236734